CLINICAL TRIAL: NCT03359161
Title: An Open Label, Descriptive Study to Evaluate the Clinical Utility of a Novel Formulation of Furosemide Delivered Subcutaneously in Patients Presenting With Early Signs of Fluid Overload
Brief Title: Clinical Utility of Subcutaneous Furosemide in Patients Presenting With Early Signs of Fluid Overload
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Development of first generation device discontinued.
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinical Protocol Version 4.0
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
Keywords: ambulatory; Subcutaneous; furosemide
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, descriptive two-phase study to evaluate the clinical effectiveness of a novel formulation of furosemide delivered by subcutaneous administration. Participants with mild to moderate signs of fluid overload will be included in the study. The study involves at home treatment with a novel formulation of subcutaneous furosemide. In the Pilot Phase (20 patients) will undergo 3 days of at home treatment for fluid overload. If determined to require more, will undergo an extra 4 days of treatment. The Investigator and her team will review the results for the first cohort and depending on the results will proceed to the Evaluation phase (40 patients).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- In-Home Subcutaneous Furosemide Treatment ARm (Experimental): Prospective, open-label arm to evaluate the clinical effectiveness of a novel formulation of furosemide delivered by subcutaneous administration.
  Interventions: Combination Product: sc2Wear Furosemide Infusor

INTERVENTIONS:
Combination Product: sc2Wear Furosemide Infusor — Subcutaneous furosemide for the treatment of fluid overload

SUMMARY:
This study will evaluate the usefulness of the subcutaneous administration of a new Lasix formulation. 20 patients will be evaluated in the first phase (pilot phase) and depending on the results, an additional 40 patients will be enrolled (Evaluation Phase). Patients with mild to moderate evidence of fluid overload who present to the cardiology service at St Elizabeth's Medical Center, Brighton, Massachusetts (SEMC) will be included in the study. Patients who qualify for thus study will be sent home with the sc2Wear™ Furosemide Infusor therapy for three days. This is a pump that patients place on their abdomen and it then delivers furosemide to the skin. Participants will be visited at home by a visiting nurse who will give them further teaching on the sc2Wear™ Furosemide Infusor. The visiting nurse will also be responsible for obtaining history (symptoms), physical examination (including inspecting the skin for adverse reactions related to the pump), and laboratory draws, supplementation of electrolytes as needed. Patients will be evaluated by the cardiology service of SEMC within 24 hours of the last dose of the sc2Wear™ Furosemide Infusor. If a patient is found to have satisfactorily responded but requires more therapy, an additional 4 days may be prescribed for total of seven consecutive treatments. If additional units are prescribed, patients will be evaluated by the cardiology service of SEMC within 24 hours of the last dose of the sc2Wear™ Furosemide infusion. Also an additionally, up to three-sc2Wear furosemide at home treatments may be used as authorized by the treating physician in case the patient experiences worsening heart failure within 30-days of enrollment (Rescue Treatment). Participants will be seen in clinic for follow up at 30±3 days after the start of the study for a post treatment.

DETAILED DESCRIPTION:
Investigational Product: Furosemide Injection, 8 mg/mL, (total dose =80 mg) administered subcutaneously by the sc2Wear Furosemide Infusor using a biphasic profile with 30 mg over the first hour and then as 12.5 mg per hour over the subsequent 4 hours. Participants may be prescribed a total of 3 days initial treatment followed by an optional additional 4 days of sc2Wear furosemide treatment based on initial clinical response.

Study Objectives: 1.) Evaluate the clinical effect of sc2Wear furosemide Infusor in the in-home management of mild to moderate decompensated heart failure.

2.) Evaluate the safety and tolerability of sc2Wear furosemide Infusor in the in-home management of mild to moderate decompensated heart failure.

Screening Phase:

The cardiology service will screen patients with mild to moderate fluid overload. Patients who present with other serious or life threatening condition for which hospitalization would be indicated are excluded. Women of child bearing potential will be screened for pregnancy with a urine pregnancy test. Eligible participants will be educated on device preparation, placement, removal and care in accordance with the Instructions of Use Manual. The screening phase includes evaluation of the home situation to ascertain that sufficient support is or can be made available for at home treatment as an alternative to inpatient care. In appropriate settings, lay caregiver will also be trained.

Pilot Phase. Patients will be visited daily by Steward Home Care and Hospice for home health nursing services in accordance with standard procedures. Nursing services will include checking vitals, obtaining blood samples and evaluation for clinical improvement or worsening. The first visit will be performed within 24 hours after enrollment.

Study Procedures: The first sc2Wear Infusor will be prepared and placed on the patient as part of the training. The patient will go home with the sc2Wear furosemide Infusor in place on the abdomen to be activated upon arrival at home. Participants will be treated with the sc2Wear furosemide Infusor daily for 3 consecutive days at home. Participants will be evaluated by the cardiology service of SEMC within 24 hours after the 3rd dose of sc2Wear furosemide. If a patient was found to have responded satisfactorily but requires additional parenteral diuretics an additional 4 days may be prescribed for a total of 7 consecutive treatments. If additional units are prescribed patients are to be evaluated the cardiology service of SEMC within 24 hours after the last dose of sc2Wear furosemide Infusor. If the subject requires further parenteral diuresis after the 7 days of at home treatment, they will be converted to usual care at that time, which may require inpatient care. Participants will be instructed to record daily morning weights during and after treatment until the second post treatment evaluation. Interim clinic visits and laboratory assessments may be required based on clinical considerations.

The following parameters will be studied at Baseline and follow-up treatment visits.

* Body Weight
* Vital signs
* HF Physical examination
* Dyspnea scale
* Routine laboratory panel (incl. electrolyte, pro-BNP)
* Adverse events
* Injection site assessment Participants will visit the clinic 30 ± 3 days after the start of the study for a post treatment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Symptomatic and chronic heart failure (NYHA Class II and III).
* Patients on guideline directed medical therapy 90 days prior to enrollment.
* Adequate home environment for at-home treatment.
* Presenting or referred to the clinic because of evidence of worsening heart failure with fluid overload (decompensation).
* A modification in oral diuretics is not clinically appropriate as deemed by the investigator.
* Estimated excess fluid weight of 4 lbs. or more from euvolemic state.
* Participant able to give informed consent for participation in trial. Agreeing to sign informed consent and HIPAA authorization.
* Understanding and willing to comply with the protocols of the trial.
* Ability of the participant or caregiver to independently apply the investigational device and medication

Exclusion Criteria:

* ACC/AHA Stage D heart failure or patients requiring IV inotrope therapy.
* Massive volume overload (e.g. >20 lbs. of estimated fluid weight) or anasarca.
* Suspected high risk clinical instability with outpatient treatment.
* Pregnant females or women of child-bearing age who are not willing to use an adequate form of contraception.
* Chronic Obstructive Pulmonary Disease (COPD) moderate or worse: FEV1/FCV ratio <0.7 and FEV1 <60 percent predicted.
* Rapid atrial fibrillation (AF) (HR >100b/min)
* Hypoxia (resting O2 saturation <90%).
* Hypotension (systolic blood pressure (SBP) BP < 90 mmHg).
* Uncontrolled diabetes mellitus (DM) (admission glucose levels > 300 mg/dL).
* Advanced renal disease (eGFR < 30mL/min/1.73m2).
* Acute coronary syndrome.
* Serum potassium (K) <3.2 mmol/L or > 5.5mmol/L.
* On experimental medication or currently participating in an interventional cardiovascular research study, other than an observational or registry study.
* Having received intravenous furosemide within 24 hours prior to enrollment.
* Urinary tract abnormality or disorder interfering with urination.
* Allergy to the active and inactive ingredients of the study medication.
* Inability to comply with study requirements.
* Ongoing substance abuse.
* Concern that the current episode of decompensation was precipitated by a serious medical condition which may require additional evaluation or treatment.
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Tsao, MD, Principal Investigator — St. Elizabeth's Medical Center
Locations (1):
- St ELizabeth's Medical Center, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Started | 9
Pilot Phase (Pilot Phase) | 9
Completed | 9 (Prematurely terminated after 9 patients.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Weight change between enrollment/screening compared to last observation
Time Frame: 30 days
Measure: Median (Full Range); unit: pounds
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
pounds | -3 [-7 to 6.5]

2. Primary Outcome: Pro BNP Change
Description: Reduction in pro-BNP between enrollment/screening compared to last observation
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
pg/ml | 412.9 (0)

3. Primary Outcome: Survival
Description: % of patients alive 30 days post enrollment
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
percentage of participants | 100

4. Primary Outcome: Hospital Admission for Heart Failure
Description: % of patients without hospitalization for worsening HF within 30 days after enrollment
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
percentage of participants | 89

5. Primary Outcome: Heart Failure Related Events
Description: % of patients without a significant Heart Failure related medical events within 30 days after enrollment.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
percentage of participants | 100

6. Primary Outcome: Extra Furosemide Treatment
Description: Percentage of patients requiring additional 4 days of diuresis
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
Participants | 6

7. Primary Outcome: Number of Participants That Discontinued Due to Presence of Skin Reaction to Drug or Device/Adhesive
Description: The number of participants that discontinued study participation due to the presence of a skin reaction to the drug or device/adhesive.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | In-Home Subcutaneous Furosemide Treatment ARm
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT03359161/Prot_SAP_000.pdf